CLINICAL TRIAL: NCT05710601
Title: Effects of Tissue Sealers on Minor Laparoscopic Procedures Between Obstetrics and Gynecology Residents
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Gaetano Riemma, Primary Investigator, University of Campania Luigi Vanvitelli
Other Study IDs: 712-15-11-19
Record Dates: First submitted 2023-01-14; First posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Benign Gynecologic Neoplasm
MeSH Terms: interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tissue sealers: Procedures performed using a 5 mm diameter, 35 cm length curved branch radiofrequency tissue sealer connected to a dedicated electric generator
  Interventions: Procedure: Laparoscopy
- Bipolar forceps: Procedures performed using a 5 mm diameter, 35 cm classic rotating bipolar forceps
  Interventions: Procedure: Laparoscopy

INTERVENTIONS:
Procedure: Laparoscopy — Operative laparoscopies carried out according to the most recent national guidelines and following the good clinical practice of our operative unit.

SUMMARY:
The kind of equipment used during laparoscopic surgery may have an effect on how quickly resident surgeons improve their skills.

The effects of these technologies on various general and specialized procedures have been the subject of numerous research, all of which have produced comparable results in terms of efficacy and safety. Although a minimally invasive laparoscopy represents the gold standard method in over 70% of procedures for uterine and adnexal benign diseases, there is a paucity of evidence regarding the potential advantages or disadvantages of such kinds of devices in gynecologic laparoscopy.

Based on this, the purpose of this study was to determine whether using a hemostatic surgical device affects how quickly gynecology residents learn to execute simple laparoscopic procedures and how well they perform surgically.

ELIGIBILITY:
Inclusion Criteria:

* Senior gynecological surgeons
* At least 4 years of residency in gynecology

Exclusion Criteria:

* Junior residents, fellows, consultants
* Operative procedures due to malignancy
* Women who were not suitable for or denied a laparoscopic approach
* Declined the procedure
* Did not sign a written informed consent form
* Suffering from a gynecologic malignant disease or severe systemic illnesses
* Laparotomic conversion

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients referred from the outpatient gynecological clinics of our unit who, according to national and international treatment guidelines, were eligible for a planned laparoscopic surgery.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Vision of the surgical field | 7 days
  Numeric Rate Scale (NRS) 0-10 considering 0 for "inadequate vision" and 10 for "optimal vision"
Interpretation of the difficulty of the intervention | 7 days
  NRS 0-10 (considering 0 for "extremely easy" and 10 for "extremely difficult")

SECONDARY OUTCOMES:
Overall procedural satisfaction | 7 days
  NRS 0-10 (considering 0 for "complicated or incomplete procedure" and 10 for "uncomplicated and satisfying intervention")
Procedure time | Procedure

CONTACTS AND LOCATIONS:
Locations (1):
- University of Campania Luigi Vanvitelli, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No